CLINICAL TRIAL: NCT07178730
Title: NeoAdjuvant Dynamic Marker - Adjusted Personalized Therapy Comparing Sacituzumab Govitecan+Pembrolizumab vs. SoC Chemotherapy in Clinical Stage II-III, Triple-negative Early Breast Cancer
Brief Title: NeoAdjuvant Therapy Comparing Sacituzumab Govitecan+Pembrolizumab vs. SoC Chemotherapy in Clinical Stage II-III, Triple-negative Early Breast Cancer
Acronym: ADAPT-TN-IV
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM15 (ADAPT-TN-IV); 2024-516734-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a multicentre, interventional, prospective, two-cohort, two-arm, partially randomized, open-label, controlled neoadjuvant, phase III trial evaluating the efficacy and safety of SG+PEM vs. SoC in stage II-III early TNBC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort I (non-randomized) (Other): Cohort I will include patients with clinical stage II disease at baseline who have a cCR after up to 12 weeks of NACT with CARBO/PAC and PEM.
  After surgery, patients with a pCR (ypT0/is, ypN0) will not receive further chemotherapy (CTx) but continue on SoC treatment according to current valid treatment guidelines for breast cancer at investigator´s discretion.
  Patients with residual disease should be considered for postoperative SoC treatment, which may include further CTx (e.g., AC/EC x 4, q2w or q3w or Capecitabine) plus PEM or Olaparib (in patients with gBRCA mutations) according to current valid treatment guidelines for breast cancer and per investigator´s discretion.
  Interventions: Drug: SoC Chemotherapy
- Cohort II (randomized) - Sacituzumab govitecan + pembrolizumab (SG+PEM) (Experimental): neoadjuvant SG+PEM (4 cycles), followed by surgery and pCR-dependent post-neoadjuvant SoC treatment according to current valid treatment guidelines for breast cancer and per investigator´s discretion.
  Interventions: Drug: Sacituzumab govitecan; Drug: Pembrolizumab 25 mg/1 ML Intravenous Solution [KEYTRUDA]
- Cohort II (randomized) - Standard-of-care chemotherapy + pembrolizumab (SoC CTx+PEM) (Active Comparator): SoC, e.g., AC x 4 + PEM or EC x 4 + PEM, followed by surgery and pCR-dependent post-neoadjuvant SoC treatment, e.g., AC x 4 * PEM or EC x 4 + PEM, or Capecitabine + PEM or Olaparib (in patients with gBRCA mutations), according to current valid treatment guidelines for breast cancer and per investigator´s discretion.
  Interventions: Drug: Pembrolizumab 25 mg/1 ML Intravenous Solution [KEYTRUDA]; Drug: SoC Chemotherapy

INTERVENTIONS:
Drug: Sacituzumab govitecan — SG is administered at 10 mg/kg as an intravenous (i.v.) infusion on Days 1 and 8 of a 21-day cycle.
  The dose of SG will be calculated based on actual weight at randomization (using weight obtained either at enrolment or on Cycle 1 Day 1) and remains constant throughout the study, unless there is a > 10% change in body weight from baseline. Modifications to the study drug doses administered should be made for a > 10% change in body weight from baseline and according to local and regional prescribing standards. Dose modifications for changes in body weight < 10% may be made according to local institutional guidelines.
  SG is administered via i.v. infusion as described below with additional information available in the current version of the SmPC.
  Other Names: Trodelvy
  Arms: Cohort II (randomized) - Sacituzumab govitecan + pembrolizumab (SG+PEM)
Drug: Pembrolizumab 25 mg/1 ML Intravenous Solution [KEYTRUDA] — Pembrolizumab 200 mg will be administered as a 30-minute i.v. infusion every 3 weeks.
  Other Names: Keytruda
  Arms: Cohort II (randomized) - Sacituzumab govitecan + pembrolizumab (SG+PEM); Cohort II (randomized) - Standard-of-care chemotherapy + pembrolizumab (SoC CTx+PEM)
Drug: SoC Chemotherapy — Standard of care chemotherapy as per common treatment guidelines and recommendations
  Other Names: diverse
  Arms: Cohort I (non-randomized); Cohort II (randomized) - Standard-of-care chemotherapy + pembrolizumab (SoC CTx+PEM)

SUMMARY:
TNBC is a heterogeneous disease with distinct pathological, genetic, and clinical features among subtypes. Treatment results for high-risk primary TNBC remain poor compared to other breast cancer subtypes. Preoperative chemotherapy is the standard of care for patients with stage II or III primary TNBC. Multiple lines of clinical evidence demonstrate that TNBC patients who achieve a pCR to NACT, (ypT0/is ypN0), have an excellent long-term prognosis. A meta-analysis of individual patient data confirmed a strong association of pCR after NACT with improved long-term event-free survival (EFS, hazard ratio [HR] 0.24) and overall survival (OS, HR 0.16) benefit. Taxane- and anthracycline-based neoadjuvant regimens generally result in pCR rates between 25-50% [REFs], whereas the addition of platinum increases pCR rates to approximately 50-55%.

The KEYNOTE-522 trial has demonstrated that the addition of the immune-checkpoint inhibitor PEM to anthracycline- (AC), taxane- and platinum-based NACT resulted in a significant increase in pCR rates to nearly 65%, associated with a significant reduction of recurrences (EFS, HR 0.65 at 5 years) and improvement of OS (HR 0.66). Based on these results, the KEYNOTE-522 regimen has been approved by the FDA and EMA and has become the standard of care for patients with stage II or III TNBC.

Despite this significant progress, two major questions remain unresolved which will be investigated in the ADAPT-TN-IV trial:

1. Do all patients require the full 6 months of NACT as per KEYNOTE-522 or is there a subgroup of patients who are sufficiently treated with 12 weeks of NACT plus PEM?
2. Can incorporation of ADCs into the KEYNOTE-522 regimen improve response and outcomes in patients without an optimal early response? The outcome of patients with residual disease after 24 weeks of NACT and PEM remains suboptimal and there is an urgent need for more effective strategies. ADCs such as SG have demonstrated superior efficacy compared to standard chemotherapy in metastatic TNBC, resulting in substantially higher response rates and improved progression-free (PFS) and OS. Combination studies of ADCs and immunotherapy in metastatic TNBC have demonstrated significant activity, suggesting possible synergistic activity It is therefore a logical next step to investigate, whether the incorporation of SG in the NACT regimen can improve pCR rates and EFS results in patients who have residual clinical disease after 12 weeks of NACT with CARBO/PAC + PEM.

DETAILED DESCRIPTION:
The trial will have two cohorts.

COHORT I - SoC DE-ESCALATION Cohort I will include patients with clinical stage II TNBC who have achieved a cCR to 12 weeks of NACT with CARBO/ PAC, and PEM. The trial will evaluate whether these patients can be safely spared from further chemotherapy (CTx) and directly proceed to surgery.

If it is unclear whether patients have a cCR, a tumour biopsy (by ultrasound or mammography/MRI-guided) is required to confirm that there is no evidence of residual invasive disease.

After surgery, patients with a pCR (ypT0/is, ypN0) will not receive further chemotherapy, but continue otherwise on SoC treatment.

Patients with residual disease should be considered for postoperative SoC treatment, which might include further CTx (e.g., AC or AC x4) plus PEM or OLA (in patients with gBRCA mutations).

COHORT II - ADC-INTENSIFICATION (STUDY TREATMENT) vs. SoC Cohort II will include all clinical stage III-patients and stage II patients without a cCR after 12 weeks of NACT with CARBO/ PAC and PEM.

If it is unclear whether patients have a cCR, a tumour biopsy (by ultrasound or mammography/MRI-guided) is required to confirm that there is no evidence of residual invasive disease.

These patients will be randomized 1:1 to further neoadjuvant treatment in either

* Arm 1: neoadjuvant SG+PEM, followed by surgery and pCR-dependent post-neoadjuvant SoC treatment or
* Arm 2: SoC CTx+SoC, followed by surgery and pCR-dependent post-neoadjuvant SoC treatment

ELIGIBILITY:
Inclusion Criteria:

Minimal eligibility criteria to be met for registration in the clinical trial:

1. TNBC: ER = 0%, PR = 0%, and HER2- (i.e., immunohistochemistry [IHC] with DAKO score ≤ 1 or fluorescence in situ hybridization [FISH]-negative)
2. or TNBC-like: ER ≤ 10% positive cells in IHC, PR < 10% positive cells in IHC, and HER2- (i.e., IHC with DAKO score ≤ 1 or FISH negative)
3. All patients, independent from gender
4. ≥18 years at diagnosis
5. Histologically confirmed unilateral, primary invasive carcinoma of the breast Note: bilateral, multicentric, or multifocal carcinoma may be included, if there is a clear target (primary) lesion, that is subject to treatment decisions and solely evaluated and documented for study purposes. Histological confirmation of all lesions as TNBC is mandatory.
6. Clinical stage II-III at baseline
7. No clinical evidence for distant metastasis (M0)
8. Cognitive and language skills to complete quality of life (QoL) questionnaires

   Additional eligibility criteria to be met for assignment to cohort I or II:
9. Completed 9-12 weeks of NACT with CARBO + PEM or PAC q1w + PEM q3w with the last dose of NACT given less than 2 weeks ago. Patients may also be considered if their NACT treatment was switched to nab-PAC due to intolerance to PAC.

   * Patients with progressive disease during taxane-CARBO treatment are allowed to participate in cohort II after consultation with sponsor, provided that at least 6-9 weeks of NACT with taxane-CARBO q1w and PEM q3w have been administered
   * Patients experiencing toxicities due to PEM, in case of contraindications or other medical reasons against PEM administration (with or without permanent discontinuation of PEM) can nevertheless be included, even if PEM will not be administered anymore. The number of patients starting the study without PEM is limited to 10%.
10. Tumour block available for central pathology review
11. Performance Status ECOG ≤ 1 or Karnofsky Index ≥ 80%
12. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
13. The patient must be capable of giving informed consent and be willing and able to comply with the requirements and restrictions in this protocol and accessible for treatment and follow-up
14. Laboratory requirements (female and male patients, ≤ 14 days old)

    * Neutrophils > 1.5 109/L,
    * Platelets > 100 109/L,
    * Total bilirubin < 1 x upper level of normal (ULN),
    * ASAT (sGOT) < 2.5 x ULN,
    * ALAT (sGPT) < 2.5 x ULN,
    * Creatinine ≤1.5 × ULN OR clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
15. Clinical assessments:

    - Normal Electrocardiogram (ECG) (within 42 days prior to induction treatment)
16. Negative pregnancy test (urine or serum) within ≤ 14 days prior to registration in premenopausal patients and immediate implementation of adequate contraceptive measures.

    Note: Pregnancy testing is to be repeated according to Schedule of Activities.
17. The following age-specific requirements apply:

    * Women aged <50 years will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the site.
    * Women aged ≥ 50 years will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments.
18. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential and need to discontinue HRT to allow confirmation of post-menopausal status prior to randomization/study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can participate without use of a contraceptive method.
19. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in Table 1 (see Section 4.4.2), from the time of enrolment and must agree to continue using such precautions for 7 months after the last dose of IMP. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic, or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
20. Female patients must not donate, or retrieve for their own use, ova from the time of randomization and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrolment in this study.
21. A male participant must agree to use a contraception as detailed in Appendix C of this protocol during the treatment period and for at least 7 months after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Known hypersensitivity to the compounds or incorporated substances of the IMPs
2. Prior malignancy with a disease-free survival of < 5 years, except curatively treated basalioma of the skin or pTis of the cervix uteri
3. Any history of invasive breast cancer
4. Previous or concurrent treatment with cytotoxic agents for any non-oncological reason unless clarified with sponsor
5. Concurrent treatment with other experimental drugs
6. Participation in another interventional clinical trial with or without any investigational, not marketed drug within 30 days or 5 half-lives of the respective drug, whichever is longer, prior to study entry. In case of other interventional trial contact Sponsor.
7. Concurrent pregnancy: patients of childbearing potential or potentially childbearing partners of male patients must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
8. Breast feeding woman
9. Reasons indicating risk of poor compliance
10. Patients not able to consent
11. Known polyneuropathy ≥ grade 2
12. Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study including recovery from major surgery, autoimmune disease, known psychiatric/substance abuse disorders, acute cystitis, ischuria, and chronic kidney disease
13. Uncontrolled infection requiring i.v. antibiotics, antivirals, or antifungals
14. History of pneumonitis haemolytic anaemia, myocarditis, sclerosing cholangitis and exocrine pancreatic insufficiency, medical history of allogenic stem cell transplants, or solid organ transplant
15. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection. Patients should be tested for HIV prior to randomization if required by local regulations or ethics committee. Patients who test positive for HIV-antibody are excluded.
16. Active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with the following detectable viral loads will be excluded.
17. Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
18. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require an HCV antibody test at enrolment and will only require HCV RNA by quantitative PCR for confirmation of active disease.
19. Patients who received live vaccines within 30 days prior to randomization.
20. Patients who are submitted to an institution by virtue of an order of a court or a governmental authority must be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Cohort I: 3-year event-free survival (EFS) | EFS 3 years
  EFS after 36 months defined as time from registration to any invasive breast cancer event, death, or secondary malignancy (same definition as iDFS) according to STEEP 2.0 criteria [103]
Cohort II: superiority of neoadjuvant treatment with SG+PEM vs. SoC with regards to event-free survival (EFS) | EFS 3 years
  EFS after 36 months defined as time from registration to any invasive breast cancer event, death, or secondary malignancy or local progress precluding surgery in neoadjuvant treated patients
Cohort II: superiority of neoadjuvant treatment with SG+PEM vs. SoC with regards to pathological complete response (pCR) rates | EFS 3 years
  pCR defined as no invasive disease in breast and lymph nodes (ypT0/is, ypN0) in patients of both arms

SECONDARY OUTCOMES:
clinical response after 12 weeks of neoadjuvant chemotherapy treatment (NACT) | 12 weeks NACT
  Clinical response measured by tumour size in mm by palpation, ultrasound, mammography, or MRI
distant disease-free survival (dDFS) | 3 years
  distant disease-free survival (dDFS)
relapse-free survival (RFS) | 3 years
  relapse-free survival (RFS)
locoregional relapse-free survival (LRFS) | 3 years
  locoregional relapse-free survival (LRFS)
overall survival (OS) | 3 years
  OS defined as time from first diagnosis to death
Health-related quality of life (HRQoL) via questionnaires EORTC-QLQ-C30, version 3.0, | Cohort I: end of the neoadjuvant treatment, at clinical response assessment, at surgery, at start of post-neoadjuvant treatment, at cycle 3, at cycle 5, at end of post-neoadjuvant treatment, 3-monthly during follow-up
  Change of Health-related quality of life (HRQoL)between baseline, after completion of SoC neoadjuvant treatment, and on following defined timepoints:
Health-related quality of life (HRQoL)via questionnaires EORTC QLQ-BR42 | Cohort I: end of the neoadjuvant treatment, at clinical response assessment, at surgery, at start of post-neoadjuvant treatment, at cycle 3, at cycle 5, at end of post-neoadjuvant treatment, 3-monthly during follow-up
  Change of Health-related quality of life (HRQoL)between baseline, after completion of SoC neoadjuvant treatment, and on following defined timepoints:
Health-related quality of life (HRQoL)via CANKADO active | Cohort I: end of the neoadjuvant treatment, at clinical response assessment, at surgery, at start of post-neoadjuvant treatment, at cycle 3, at cycle 5, at end of post-neoadjuvant treatment, 3-monthly during follow-up
  Change of Health-related quality of life (HRQoL)between baseline, after completion of SoC neoadjuvant treatment, and on following defined timepoints:
Health-related quality of life (HRQoL)via questionnaires EORTC-QLQ-C30, version 3.0, | Cohort II: end of the neoadjuvant treatment, at clinical response assessment, at cycle 3 of prolonged neoadjuvant treatment, at surgery, at start of post-neoadjuvant treatment, 3-monthly during follow-up
  Change of Health-related quality of life (HRQoL)between baseline, after completion of SoC neoadjuvant treatment, and on following defined timepoints:
HRQoL via questionnaires EORTC QLQ-BR42 | Cohort II: end of the neoadjuvant treatment, at clinical response assessment, at cycle 3 of prolonged neoadjuvant treatment, at surgery, at start of post-neoadjuvant treatment, 3-monthly during follow-up
  Change of HRQoL between baseline, after completion of SoC neoadjuvant treatment, and on following defined timepoints:
HRQoL via CANKADO active | Cohort II: end of the neoadjuvant treatment, at clinical response assessment, at cycle 3 of prolonged neoadjuvant treatment, at surgery, at start of post-neoadjuvant treatment, 3-monthly during follow-up
  Change of HRQoL between baseline, after completion of SoC neoadjuvant treatment, and on following defined timepoints:

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, PHD Dr, Principal Investigator — Westdeutsche Studiengruppe GmbH; Nadia Harbeck, Prof Dr, Principal Investigator — Breast Centre, Dept. Obstetrics & Gynaecology and CCC Munich LMU University Hospital Munich Germany; Oleg Gluz, Prof Dr, Principal Investigator — Breast Centre, Evang. Bethesda-Hospital Moenchengladbach Germany; Sherko Kuemmel, Prof Dr, Principal Investigator — Breast Centre, Kliniken Essen Mitte Essen Germany; Monika Graeser, PD Dr, Principal Investigator — Breast Centre, Marien-Hospital Witten Germany

IPD SHARING:
Plan to Share IPD: No